CLINICAL TRIAL: NCT06630689
Title: Effects of Oil and Dry Neonatal Massage on Hyperbilirubinemia and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: meral güven (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, meral güven, research assistant, Igdir University
Organization: Igdir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IU-SBF-MG-01
Record Dates: First submitted 2024-10-05; First posted 2024-10-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: hyperbilirubinemia; massage; comfort; newborn
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Intervention Model Description: The study consisted of 3 groups: control group, dry whole body massage group and oily whole body massage group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the study participants were newborns, the participants were naturally blinded to the study. Due to the nature of the study, the researcher who applied the nursing intervention to the experimental groups could not be blinded to which group the babies were assigned to. However, blinding was done for the other researchers and the statistical process in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Babies in the control group will receive treatment and care according to neonatal intensive care unit procedures. No intervention will be applied.
- Dry Full Body Massage Group (Experimental): Unlike the control group, dry whole body massage was applied to the babies who were followed up after completing the phototherapy treatment process.
  Interventions: Other: Dry Full Body Massage
- Oil Full Body Massage Group (Experimental): Unlike the control group, the babies in this group received a full body oil massage. The full body oil massage was applied using pure baby olive oil.
  Interventions: Other: Oil Full Body Massage

INTERVENTIONS:
Other: Dry Full Body Massage — Applying massage after phototherapy
  Arms: Dry Full Body Massage Group
Other: Oil Full Body Massage — Oil Full Body Massage
  Arms: Oil Full Body Massage Group

SUMMARY:
The need for infant massage may come to the forefront as a part of routine care in the neonatal intensive care unit to reduce high bilirubin levels in newborns and to reduce the need for phototherapy treatment. This study was planned to investigate the effects of oily and dry neonatal massage on hyperbilirubinemia and comfort.

DETAILED DESCRIPTION:
Hyperbilirubinemia is a common disease affecting newborns. It is a self-limiting condition, but if not properly monitored and managed, it can cause permanent neurological disorders. Hyperbilirubinemia affects approximately 8-11% of newborns and accounts for 75% of hospitalizations in the first weeks of life. Physiological jaundice occurs in newborns within the first 24-72 hours after birth; it is at its highest level on days 3-4, begins to decrease on days 5-7 and disappears completely on days 10-14, and in premature babies, it occurs after 48 hours and can take up to 4 weeks to completely resolve. Jaundice that occurs within the first 24 hours is pathological jaundice. High bilirubin levels can cause kernicterus, which can lead to serious neurological damage if not diagnosed and treated early. This condition has a 75% probability of death in infants and can cause neurological sequelae in 80% of survivors. Different treatment methods are used to reduce bilirubin levels. Frequently used methods are; exchange transfusion, phototherapy and drug therapy. Phototherapy is one of the most frequently used methods in the treatment of hyperbilirubinemia. Phototherapy has many complications such as damage to the retina and reproductive organs, dehydration in the body, skin rashes, watery stools and bronze baby syndrome. Recently, research has been conducted on different treatment approaches and new applications to manage neonatal hyperbilirubinemia and shorten the hospitalization period. It has been stated that massage and bath applications reduce bilirubin levels in newborns. Massage is the systematic manual stimulation of the soft tissues of the body with movements such as friction, pressing, rolling and touching for therapeutic purposes. Massage, which is one of the oldest healing applications and can be easily applied together with traditional treatments, is the most natural and instinctive tools.Massage in newborns is accepted as a new care method with positive effects.Neonatal massage is not a mechanical routine, but a simple, cheap and effective technique to support newborn development and to ensure that parents establish eye contact with their babies. Massage is a new, easy to apply and alternative method that can be used to reduce bilirubin levels in newborns. Baby massage can help to remove bilirubin from the body by increasing lymph and blood circulation. Massage stimulates bowel movements and causes early defecation. Increased intestinal peristalsis reduces the enterohepatic circulation of bilirubin and accelerates its excretion from the body. Studies have shown that massage significantly increases the frequency of defecation in babies. Baby massage can significantly increase the number of stools by significantly increasing the intestinal stimulation of babies with vagal activity and thus help to remove bilirubin from the body. In the findings of many studies; it has been reported that baby massage is a method that helps to remove bilirubin from the body.

ELIGIBILITY:
Inclusion Criteria:

* Being a term (37-42 weeks) newborn.
* The newborn's postnatal age is between 1st and 28th days
* The 1st and 5th Apgar score is between 7-10
* The newborn is fed orally
* The newborn's birth weight is 2500 grams and above
* Phototherapy treatment is terminated and followed up
* Receiving nutritional support for hyperbilirubinemia
* No health problems other than hyperbilirubinemia
* Stable general health status
* Parents' willingness and volunteering to participate in the study constitute the inclusion criteria for the study.

Exclusion Criteria:

-

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Newborn Comfort Behavior Scale (COMFORTneo) | 9 months
  The Newborn Comfort Behavior Scale, developed to determine sedation, need for comfort, pain or distress in infants followed in the NICU, is a five-point Likert-type scale. The five-point Likert-type scale consists of six parameters including alertness, calmness/agitation, respiratory response, crying, body movements, facial tension and muscle tone. In infants receiving mechanical ventilation, the "Respiratory Response" element is taken into account, and in those not receiving mechanical ventilation, the "Crying" element is taken into account.
Numerical Assessment Scales | 9 months
  Numerical Assessment Scales are based on the observation of the researcher. Each item in the scale is scored from 1 to 5 and evaluated over a total score. The lowest score on the scale should be 6 and the highest score should be 30. If the total score obtained from the scale is between 9-13, it means that the newborn is comfortable, and if it is between 14-30, it means that the newborn is in pain or distress and therefore not comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: meral güven, Principal Investigator — Igdir University
Locations (1):
- Igdir University, Iğdır, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't prefer